CLINICAL TRIAL: NCT01964573
Title: A Single-site, Randomized, Double-blind, Placebo-controlled, Repeated-dose Trial to Evaluate the Pharmacokinetics, Safety, and Tolerability of Rotigotine in 2 Different Dosages (2 mg / 24 Hours [10 cm2], 4 mg / 24 Hours [20 cm2]) in Healthy Korean Subjects
Brief Title: Trial to Evaluate the Pharmacokinetics, Safety, and Tolerability of Rotigotine in Healthy Korean Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SP0885
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2013-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Rotigotine; Pharmacokinetics; Healthy subjects
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine group (Experimental)
  Interventions: Drug: Rotigotine
- Placebo group (Placebo Comparator): Placebo matched to rotigotine will be administered in the same way as within the Rotigotine group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rotigotine — Day 1-3: 2 mg patch once daily
  Day 4-6: 4 mg patch once daily
  Other Names: Neupro
  Arms: Rotigotine group
Other: Placebo — Placebo patches matching with Rotigotine 2 mg patches and 4 mg patches.
  Frequency:
  Day 1-3: 2 mg patch once daily
  Day 4-6: 4 mg patch once daily
  Arms: Placebo group

SUMMARY:
The objective of this trial is to investigate the PK (Pharmacokinetic) of repeated-dose applications of the Rotigotine transdermal patch in healthy young male and female Korean subjects to be submitted to MFDS for new drug application approval.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and aged between 19 and 45 years of age (inclusive)
* Subject is healthy (no clinically relevant findings in any of the investigations of the pre-examination) as judged by the investigator
* Subject is of normal body weight as determined by a Body Mass Index (BMI) between 18 and 28 kg / m²
* Subject is Korean (both parents are pure Korean)

Exclusion Criteria:

* Subject has had a history of drug or alcohol abuse within the last 2 years
* Subject has had a history of transient ischemic attack or stroke within the last 12 months
* Subject has a history or current condition of Epilepsy and / or seizures
* Subject has a history of significant skin hypersensitivity to adhesives or other transdermal products or recently unsolved Contact Dermatitis
* Subject has a history or present condition of an Atopic or Eczematous Dermatitis, Psoriasis, and / or an active skin disease
* Female subject is pregnant or lactating
* Subject has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this trial
* Subject has a QTcB (according to Bazett´s formula) interval of ≥ 450 ms for female or ≥ 430 ms for male or any other clinically relevant Electrocardiogram (ECG) finding
* Subject has any clinically relevant abnormality in the physical examination, or any clinically relevant deviation from the normal range in the clinical chemistry, hematology, or urinalysis
* Subject has a relevant hepatic dysfunction (total Bilirubin > 2 mg /dL or Alanine Aminotransferase [ALT] or Aspartate Aminotransferase [AST] greater than 2 times the upper limit of the normal reference range)
* Subject has a positive test for Human Immunodeficiency Virus antibodies (HIV)-1/2Ab, Hepatitis B surface Antigen (HBsAg) or Hepatitis C Virus Antibody (HCV-Ab)
* Subject has a positive test for alcohol or drugs
* Subject consumes more than 150 g of alcohol / week
* Subject has made a blood donation or had a comparable blood loss (> 400 ml) within the last 3 months
* Subject smokes more than 5 cigarettes per day or has done so within previous 6 months
* Subject has a clinically relevant allergy
* Subject is taking any medication (excluding oral hormonal contraceptive) currently or within 2 weeks prior to the first day of dosing (with the exception of Acetaminophen [up to 1000 mg per day per os] which may have been taken up to 48 hours prior to commencement of dosing)
* Female subject is currently taking an oral hormonal contraceptive but less than 2 months
* Subject has a symptomatic orthostatic hypotension with a decrease of Blood Pressure (BP) from supine to standing position of ≥ 20 mmHg in systolic BP or of ≥ 10 mmHg in diastolic BP after 1 and / or 3 minutes
* Subject has a pulse rate at rest less than 45 beats per minute or more than 100 beats per minute (measured in supine position)
* Subject has a systolic Blood Pressure (BP) lower than 100 mmHg or higher than 150 mmHg or diastolic BP higher than 95 mmHg (measured in supine position)
* Subject has a current or a history of clinically relevant motor disturbance, impairment of memory, sleep disturbance or neurodegenerative disease (e.g. , Alzheimer Dementia, Diffuse, Lewy Body Dementia, Amyotrophic Lateral Sclerosis [ALS], Multiple Sclerosis)
* Subject has taken herbal medicine therapy within the last 2 weeks
* Subject consumes more than 3 cups (more than 450 ml) of caffeinated beverages per day within the last 2 weeks

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Plasma concentrations of total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Area under the plasma concentration-time curve from 0 to 24 hours at steady-state (AUC (0-24), ss) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Area under the plasma concentration-time curve from 0 to 24 hours at steady-state (AUC (0-24), ss) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Area under the plasma concentration-time curve from 0 to 24 hours at steady-state normalized by Body Weight (AUC (0-24), ss, norm (BW)) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Area under the plasma concentration-time curve from 0 to 24 hours at steady-state normalized by Body Weight (AUC (0-24), ss, norm (BW)) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Maximum plasma concentration (Cmax) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Maximum plasma concentration (Cmax) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Maximum plasma concentration normalized by Body Weight (Cmax, norm (BW)) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Maximum plasma concentration normalized by Body Weight (Cmax, norm (BW)) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from 0 to 24 hours at steady-state normalized by apparent-dose (AUC (0-24), ss, norm (apparent-dose)) of unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Area under the plasma concentration-time curve from 0 to 24 hours at steady-state normalized by apparent-dose (AUC (0-24), ss, norm (apparent-dose)) of total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Maximum plasma concentration normalized by apparent-dose (Cmax, norm (apparent-dose)) of unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Maximum plasma concentration normalized by apparent-dose (Cmax, norm (apparent-dose)) of total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Area under the plasma concentration-time curve from 0 to 24 hours at steady-state normalized by drug content (AUC (0-24), ss, norm (mgdc)) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Area under the plasma concentration-time curve from 0 to 24 hours at steady-state normalized by drug content (AUC (0-24), ss, norm (mgdc)) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Maximum plasma concentration normalized by drug content of patch (Cmax, norm (mgdc)) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Maximum plasma concentration normalized by drug content of patch (Cmax, norm (mgdc)) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Terminal half-life (t ½) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Terminal half-life (t ½) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Time to reach maximum plasma concentration during a dosing interval at steady-state (t max, ss) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Time to reach maximum plasma concentration during a dosing interval at steady-state (t max, ss) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Apparent total body clearance (CL/f) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Apparent total body clearance (CL/f) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Apparent total body clearance normalized by Body Weight (CL/f norm (BW)) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Apparent total body clearance normalized by Body Weight (CL/f norm (BW)) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Apparent total body clearance normalized by apparent-dose (CL/f norm (apparent-dose)) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Apparent total body clearance normalized by apparent-dose (CL/f norm (apparent-dose)) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Apparent volume of distribution (Vz/f) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Apparent volume of distribution (Vz/f) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Apparent volume of distribution normalized by Body Weight (Vz/f norm (BW)) for unconjugated Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Apparent volume of distribution normalized by Body Weight (Vz/f norm (BW)) for total Rotigotine | Day 3 and Day 6 predose, and 1, 2, 3, 4, 6, 8, 12, 16, 24 hours after patch application at Day 3 and 6 and 25, 26, 28, 30, 33 and 36, 48, 60, 72 hours after patch application on Day 6
Plasma concentration at steady-state directly before patch removal (C (24), ss) for total Despropyl Rotigotine | Directly before patch removal at Day 2 to Day 7
Plasma concentration at steady-state directly before patch removal (C (24), ss) for total Desthienyl Rotigotine | Directly before patch removal at Day 2 to Day 7
Plasma concentration at steady-state 30 hours after last patch application (C (30 h), ss) for total Despropyl Rotigotine | At day 7 at 30 hours after last patch application
Plasma concentration at steady-state 30 hours after last patch application (C (30 h), ss) for total Desthienyl Rotigotine | At day 7 at 30 hours after last patch application
Amount excreted into urine from 0 to 24 hours at steady-state (Ae (0-24), ss) for unconjungated Rotigotine | Day 3 and Day 6 from 0 to after 24 hours of patch application
Amount excreted into urine from 0 to 24 hours at steady-state (Ae (0-24), ss) for total Rotigotine | Day 3 and Day 6 from 0 to after 24 hours of patch application
Amount excreted into urine from 0 to 24 hours at steady-state (Ae (0-24), ss) for total Despropyl Rotigotine | Day 3 and Day 6 from 0 to after 24 hours of patch application
Amount excreted into urine from 0 to 24 hours at steady-state (Ae (0-24), ss) for total Desthienyl Rotigotine | Day 3 and Day 6 from 0 to after 24 hours of patch application
Renal Clearance (CLR) for unconjugated Rotigotine | Day 3 and Day 6 from 0 to after 24 hours of patch application
Renal Clearance (CLR) for total Rotigotine | Day 3 and Day 6 from 0 to after 24 hours of patch application

CONTACTS AND LOCATIONS:
Overall Officials: UCB, Inc., Study Director — +1 877 822 9493
Locations (1):
- Seoul, South Korea

REFERENCES:
- [Derived] Kim BH, Yu KS, Jang IJ, Soo Lim K, Kim JR, Elshoff JP, Andreas JO, Braun M, Cawello W. Pharmacokinetic properties and tolerability of rotigotine transdermal patch after repeated-dose application in healthy korean volunteers. Clin Ther. 2015 Apr 1;37(4):902-12. doi: 10.1016/j.clinthera.2015.01.013. Epub 2015 Mar 16. PMID 25791613